CLINICAL TRIAL: NCT07028424
Title: Pancreatic Cancer First-line NALIRIFOX Optimization With 5-FU Maintenance and Role of Antibiotics and Microbiota Exploration in Second-line Treatment - A Non-comparative, Randomized Phase II PANORAMIX GERCOR G-116 PRODIGE 105 Study.
Brief Title: PANORAMIX : Optimizing 1st-line NALIRIFOX and Exploring Microbiota's Role in 2nd Line Pancreatic Cancer Treatment
Acronym: PANORAMIX
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Collaborators: Servier (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PANORAMIX G-116 PRODIGE 105
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: PDAC - Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — irinotecan sucrosofate; Ciprofloxacin; Paclitaxel; Gemcitabine; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Intervention Model Description: This is a randomized, non-comparative two-step study in patients with metastatic PDAC.
  STEP 1 (main objective) This is a two-arm, open-label, randomized (2:1), non-comparative single stage phase II study to assess the efficacy of 5-FU-based maintenance after NALIRIFOX initiation (Arm 1A) versus standard NALIRIFOX in patients with metastatic PDAC (Arm 1B).
  STEP 2 (secondary exploratory objective) This is a two-arm, double-blinded, randomized (1:1), non-comparative, two-stage phase II with ciprofloxacin + gemcitabine-based chemotherapy (gemcitabine +/- paclitaxel) regimen (Arm 2A) versus gemcitabine-based chemotherapy (gemcitabine +/- paclitaxel) regimen + placebo (Arm 2B)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only STEP 2 of the study is masked; a double-blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- STEP 1 - Experimental Arm 1A : First-line NALIRIFOX with LV5FU2 [5-FU/leucovorin] maintenance) (Experimental): NALIRIFOX (NAL-IRI + 5FU/LV + oxaliplatin; 8 cycles) followed by LV5FU2 maintenance administered every 14 days (2 weeks) followed by NALIRIFOX reintroduction (for maximum 8 cycles) followed by LV5FU2 maintenance
  Interventions: Drug: Nal-IRI; Drug: Oxaliplatin; Drug: Leucovorin; Drug: 5-Fluorouracil
- STEP 1 - Arm 1B: NALIRIFOX (Active Comparator): NALIRIFOX until disease progression or unacceptable toxicity
  Interventions: Drug: Nal-IRI; Drug: Oxaliplatin; Drug: Leucovorin; Drug: 5-Fluorouracil
- STEP 2 - Arm 2A: Gemcitabine +/- paclitaxel + ciprofloxacin (Experimental): Gemcitabine: 1,000 mg/m2 intravenously (IV) over 30 minutes weekly on days 1, 8, 15 of each 28-days cycle.
  +/- Paclitaxel 80 mg/m2 weekly on days 1, 8, 15 of each 28-days cycle (at the discretion of investigator).
  Ciprofloxacin (6 capsules/cycle, withhold if gemcitabine is not administered): 500 mg twice daily (morning and evening; 12 hours should elapse between two doses) on days 1, 8, 15 (on day of gemcitabine infusion) for a maximum of 6 months.
  Interventions: Drug: Ciprofloxacin; Drug: Paclitaxel; Drug: Gemcitabine
- STEP 2 - Arm 2B: Gemcitabine +/- paclitaxel + placebo (Active Comparator): Gemcitabine: 1,000 mg/m2 intravenously (IV) over 30 minutes weekly on days 1, 8, 15 of each 28-days cycle.
  +/- Paclitaxel 80 mg/m2 weekly on days 1, 8, 15 of each 28-days cycle (at the discretion of investigator).
  Placebo (6 capsules/cycle, withhold if gemcitabine is not administered): 500 mg twice daily (morning and evening; 12 hours should elapse between two doses) on days 1, 8, 15 (on day of gemcitabine infusion) for a maximum of 6 months.
  Interventions: Drug: Paclitaxel; Drug: Gemcitabine; Other: Placebo

INTERVENTIONS:
Drug: Nal-IRI — NAL-IRI 50 mg/m2, administered over 80-100 minutes, on day 1 of a 14-days cycle
  Other Names: iposomal irinotecan
  Arms: STEP 1 - Arm 1B: NALIRIFOX; STEP 1 - Experimental Arm 1A : First-line NALIRIFOX with LV5FU2 [5-FU/leucovorin] maintenance)
Drug: Ciprofloxacin — 6 capsules/cycle : 500 mg twice daily on days 1, 8, 15 (on day of gemcitabine infusion) for a maximum of 6 months
  Arms: STEP 2 - Arm 2A: Gemcitabine +/- paclitaxel + ciprofloxacin
Drug: Paclitaxel — 80 mg/m2 weekly on days 1, 8, 15 of each 28-days cycle (at the discretion of investigator)
  Arms: STEP 2 - Arm 2A: Gemcitabine +/- paclitaxel + ciprofloxacin; STEP 2 - Arm 2B: Gemcitabine +/- paclitaxel + placebo
Drug: Gemcitabine — 1,000 mg/m2 intravenously (IV) over 30 minutes weekly on days 1, 8, 15 of each 28-days cycle
  Arms: STEP 2 - Arm 2A: Gemcitabine +/- paclitaxel + ciprofloxacin; STEP 2 - Arm 2B: Gemcitabine +/- paclitaxel + placebo
Drug: Oxaliplatin — 60 mg/m2 (starting 2 hours later, administered over 110-130 minutes) on day 1
  Arms: STEP 1 - Arm 1B: NALIRIFOX; STEP 1 - Experimental Arm 1A : First-line NALIRIFOX with LV5FU2 [5-FU/leucovorin] maintenance)
Drug: Leucovorin — As part of NALIRIFOX -for 8 cycle treatment: (L + D racemic form) 400 mg/m2 on day 1 (equivalent to 200 mg/m2 levoleucovorin) (starting 30 minutes after oxaliplatin, administered over 25-35 minutes)
  As part of LV5FU2 maintenance treatment: 400 mg/m2 IV infusion over 30 min on day 1 (equivalent to 200 mg/m2 levoleucovorin). LV could be administered over 2 hours to oxaliplatin according to The National Thesaurus of Digestive Oncology (TNCD) https://www.snfge.org/sites/www.snfge.org/files/tncd/2024-05/tncd_chap-09-cancer-pancre%CC%81as_2024-05-17_1.pdf, at investigator's discretion
  Arms: STEP 1 - Arm 1B: NALIRIFOX; STEP 1 - Experimental Arm 1A : First-line NALIRIFOX with LV5FU2 [5-FU/leucovorin] maintenance)
Drug: 5-Fluorouracil — As part of NALIRIFOX -for 8 cycle treatment: 2400 mg/m² IV initiated on day 1, with continuous infusion over 46 hours (no bolus infusion with 5-FU)
  As part of LV5FU2 maintenance treatment: 400 mg/m2 bolus over 10 min then 2,400 mg/m2 IV infusion over 46h
  Arms: STEP 1 - Arm 1B: NALIRIFOX; STEP 1 - Experimental Arm 1A : First-line NALIRIFOX with LV5FU2 [5-FU/leucovorin] maintenance)
Other: Placebo — 6 capsules/cycle : 500 mg twice daily (morning and evening; 12 hours should elapse between two doses) on days 1, 8, 15 (on day of gemcitabine infusion) for a maximum of 6 months
  Arms: STEP 2 - Arm 2B: Gemcitabine +/- paclitaxel + placebo

SUMMARY:
The main objective of PANORAMIX phase II trial is to optimize first-lie (L1) NALIRIFOX treatment for pancreatic cancer through the implementation of 5-fluorouracil (5-FU) maintenance therapy. Additionally, it aims to investigate the role of antibiotics and microbiota in second-line (L2) treatment.

DETAILED DESCRIPTION:
This randomized non-comparative phase II study consists of two sequential steps.

Step 1 (main objective), the primary goal is to assess the efficacy of a maintenance strategy with LV5FU2 alone after disease control with first-line NALIRIFOX-based chemotherapy in patients with metastatic pancreatic ductal adenocarcinoma (PDAC).

Step 2 of the study (exploratory objective), aim is to assess the efficacy and safety of the addition of fluoroquinolone (ciprofloxacin) to gemcitabine-based chemotherapy in second-line setting.

ELIGIBILITY:
Inclusion Criteria:

Overlapping inclusion criteria for STEP 1 AND STEP 2

1. Written informed consent obtained from the patient prior to performing any protocol-related procedures, including screening evaluations (only after interim analysis at Step 2 for patients who were not randomized in first randomization [R1]),
2. Age ≥18 years old. STEP 1: The patient over 75 years of age is eligible only if the patient's G8 score (G8 questionnaire) is > 14,
3. Eastern Cooperative Oncology Group performance status (ECOG PS) 0-1,
4. Histologically or cytologically proven PDAC,
5. ≥1 measurable lesion according to RECIST v 1.1 (Computed tomography thorax-abdomen-pelvis [TAP-CT] scan ≤ 4 weeks), Note: abdominal magnetic resonance imaging (MRI) is allowed (e.g., in case of contra-indication to CT scan contrast injection) provided that this imaging modality is used consistently throughout the tumor evaluations,
6. Availability of archival tissue samples for exploratory research. Step 2: can be the same as in Step 1 or it can be newly obtained sample,
7. Adequate organ function, obtained within 21 days prior to randomization of study treatment, as defined by the following:

   * Serum aspartate aminotransferase (AST) and serum alanine aminotransferase (ALT) ≤3 x upper limit of normal (ULN; ≤ 5 x ULN in case of liver metastases) - STEP 2, if paclitaxel administration,
   * Total serum bilirubin < 1.5 x ULN (STEP 2, if paclitaxel administration),
   * Serum albumin ≥ 28 g/L,
   * Hemoglobin ≥ 9.0 g/dl,
   * Absolute neutrophil count (ANC) ≥ 2 x 10^9L,
   * Platelets - STEP 1: ≥ 150 x 10^9L; STEP 2: ≥ 100 x 10^9L,
   * Creatinine clearance ≥ 50 mL/min (Modification of the Diet in Renal Disease [MDRD]),
8. Evidence of post-menopausal status or negative serum pregnancy test within 7 days before starting study treatment for female pre- menopausal patients. Women of childbearing potential (WOCBP) should use effective contraception during study treatment and: 1 month (paclitaxel), 6 months (5FU, LV), 7 months (NAL-IRI), 15 months (oxaliplatin), and 6 months (gemcitabine+/-paclitaxel and ciprofloxacin/placebo) after the patient's last dose of treatment. Males who are fertile should use effective contraception during study treatment and 4 months (NAL-IRI), 6 months (5-FU, LV), 12 months (oxaliplatin), and 6 months (gemcitabine+/-paclitaxel and ciprofloxacin/placebo) after the patient's last dose of treatment.
9. Willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up,
10. Registration in a National Health Care System (PUMa - Protection Universelle Maladie included).

    Distinct inclusion criteria for STEP 1 and STEP 2 STEP 1
11. No prior first-line chemotherapy (5-FU or gemcitabine based, or FOLFIRINOX) for metastatic disease; if treatment with any investigational medicinal product (IMP) the delay before the last dose and inclusion more than or equal to 28 days, Note: relapse after FOLFIRINOX adjuvant chemotherapy in case of resectable disease is NOT allowed,
12. No dihydropyrimidine dehydrogenase (DPD) deficiency (Uracilemia dosage >16 ng/ml), Uracilemia dosing results must be available before inclusion).

STEP 2 11. Metastatic disease, 12. L2 therapy after progression under 5-FU-based chemotherapy for localized/locally advanced or metastatic stage, Note: relapse <4 months after the end of adjuvant chemotherapy in case of resectable disease is allowed.

Exclusion Criteria:

Overlapping exclusion criteria for STEP 1 AND STEP 2

1. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or the follow-up period of an interventional study,
2. History of allogenic organ transplantation or active autoimmune, connective tissue disorder, or inflammatory disease requiring systemic treatment,
3. Diagnosis of any second malignancy that required any treatment within the last 3 years, except for adequately treated basal cell or squamous cell skin cancer, or in situ carcinoma of the cervix uteri,
4. History of idiopathic pulmonary fibrosis, interstitial lung disease (ILD), drug-induced pneumonitis, organizing pneumonia, or evidence of active pneumonitis on screening (TAP-CT-scan),
5. Current systemic steroid therapy (>10 mg daily dose of prednisone or equivalent; minimal wash-out of 1 week [7 days]) or immunosuppressive therapy,
6. Prior radiotherapy treatment to more than 30% of the bone marrow or a wide field of radiation within 4 weeks (30 days) prior to the first dose of study drug,
7. Major surgical procedure (as defined by the Investigator) within 4 weeks (30 days) prior to the first dose of trial treatment (Step 1 and Step 2), Note: Local surgery of isolated lesions for palliative intent is acceptable,
8. Uncontrolled central nervous system metastases and/or carcinomatous meningitis,
9. Uncontrolled massive pleural effusion or massive ascites,
10. Uncontrolled intercurrent illness, including but not limited to, symptomatic congestive heart failure or coronary disease, peripheral artery disease, severe chronic obstructive pulmonary disease, decompensated cirrhosis, serious chronic gastrointestinal conditions (e.g. bleeding, inflammation, occlusion, malabsorption syndrome, ulcerative colitis, gastrointestinal ulceration, infection or sepsis, inflammatory bowel disease or partial bowel obstruction) associated with diarrhea, or geographical/social/ psychiatric illness situations that would limit compliance with study requirement and study follow-up, substantially increase risk of incurring AEs, or compromise the ability of the patient to give written informed consent,
11. History or current evidence of any condition, therapy, laboratory abnormality that might confound the results of the trial, interfere with participation for the full duration of the trial, or is not in the best interest of the participant in the opinion of the treating investigator,
12. QT/QTc interval >470 ms (for women) and > 450 ms (for men), previous ventricular arrhythmia, known or suspected long-QT syndrome, Note: Caution is required when using medicinal products with human thymidine kinase substrates, e.g. zidovudine and other drugs known to prolong the QTc interval (exhaustive list on https: //www.crediblemeds.org.")
13. Known or suspected allergy or hypersensitivity to any of the study drugs or any of the study drug excipients,
14. Active bacterial, viral, or fungal infection requiring systemic therapy, including tuberculosis, hepatitis B (HBV, known positive HBV surface antigen [HbsAg] result), hepatitis C (HBC, with positive RNA), or human immunodeficiency virus (HIV positive 1/2 antibodies), Note: Patients with past HBV infection or resolved HBV infection (defined as having a negative HbsAg test and a positive hepatitis B core antigen [HBc] antibody test) are eligible; patients with previously treated and cured HCV infection (negative RNA) are also eligible,
15. Live vaccine administration within 4 weeks (30 days) prior to the first dose of study treatment,
16. Pregnancy/breast-feeding/lactation,
17. Under a legal protection measure (guardianship, curatorship, or judicial safeguard), administrative decision, and/or incapable of giving his/her consent.

Distinct exclusion criteria for STEP 1 and STEP 2 STEP1 18. Any unresolved NCI CTCAE toxicity of grade ≥ 2 from previous anticancer therapy (including peripheral neuropathy of grade ≥ 1) except for alopecia or vitiligo, 19. Any previous chemotherapy for advanced disease, 20. Uncontrolled central nervous system metastases and/or carcinomatous meningitis, 21. Peripheral neuropathy with functional discomfort > grade 2, 22. Clinically significant active heart disease or myocardial infarction within 6 months given the cardiotoxicity of 5-FU, 23. Abnormal values of potassium, magnesium, and calcium levels at inclusion, 24. Patients with known homozygous UGT1A1*28 (Gilbert's disease), 25. Any use of strong CYP3A4 inducers/inhibitors and/or strong UGT1A1 inhibitors (patients are ineligible if unable to discontinue the use of strong CYP3A4 or UGT1A1 inhibitors at least 1 week or strong CYP3A4 inducers at least 2 weeks prior to receiving first dose of NAL-IRI injection), or presence of any other contraindications for irinotecan), 26. Brivudine-based treatment within 4 weeks preceding treatment initiation. STEP 2 18. Antibiotics use in the month before the day of treatment initiation or for > 5 days within 3 months before the day of treatment initiation, 19. Previous gemcitabine-based chemotherapy, 20. Known previous colonization or infection with K. pneumoniae resistant to quinolones, 21. Prophylactic phenytoin within 1 week (7 days) prior to the first dose of study treatment, 22. Any contra-indication to ciprofloxacin: history of fluoroquinolone-related severe side effects (muscle, tendons, joint…), severe aortic disease (aneurysm, dissection), myasthenia, epilepsy, 23. Inability to take oral treatment, 24. Concomitant medication with CYP1A2 substrates (e.g., theophylline, clozapine, duloxetine, tizanidine, olanzapine, propranolol, amitryptilin, and methotrexate, 25. Known glucose-6-phosphate dehydrogenase deficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2029-07 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
6-month progression-free survival (PFS) rate post randomization Step 1 (R1) in Arm 1A | 6 months
  To assess the efficacy of a 6-month PFS rate post R1 in patients with metastatic PDAC who received first-line (L1) NALIRIFOX with LV5FU2 (5-FU/leucovorin) maintenance strategy during Step 1 (Arm 1A).

SECONDARY OUTCOMES:
Progression-free survival first-line (PFS-L1) post randomization Step 1 (R1) in Arm 1A and in Arm 1B | up to 5 years
  To assess PFS-L1 post R1 in Arm 1A and Arm 1B
Progression-free survival (PFS) post NALIRIFOX reintroduction (PFS-reintro) in Arm 1A | up to 5 years
  To assess PFS-reintro in Arm 1A
Overall survival post randomization Step 1 (OS-R1) in Arm 1A and in Arm 1B | up to 5 years
  To assess OS-R1 in Arm 1A and Arm 1B
Overall response rate of first-line (ORR-L1) at 4 months in Arm 1A and in Arm 1B | 4 months
  To assess ORR-L1 at 4 months in Arm 1A and Arm 1B, according to RECIST 1.1
Overall response rate post NALIRIFOX reintroduction (ORR-RI) in Arm 1A | up to 5 years
  To assess ORR-RI in Arm 1A
Best response rate of first-line (BRR-L1) in Arm 1A and in Arm 1B | up to 5 years
  To assess BRR-L1 in Arm 1A and Arm 1B
Best response rate of first-line after reintroduction of NALIRIFOX (BRR-L1R) in Arm 1A | up to 5 years
  To assess BRR-L1R in Arm 1A
Duration of disease control (DDC) in Arm 1A and in Arm 1B | up to 5 years
  To assess DDC in Arm 1A and in Arm 1B
Grade 3-4 adverse events (AEs)/serious AEs (SAEs) related to treatment | until 28 days after end of treatment visit
  To assess safety (only grade 3-4 AEs/SAEs related to treatment in Arm 1A and Arm 1B, according to the NCI CTCAE v5.0
Rate of peripheral neuropathy in Arm 1A and Arm 1B | up to 5 years
  To assess the rate of peripheral neuropathy (all grade and severe [grade 3-5] adverse events [AEs] in Arm 1A and Arm 1B, according to NCI CTCAE v5.0
Health-related quality of life (HRQoL) by EORTC QLQ-C3 in Arm 1A and in Arm 1B | up to 5 years
  To assess HRQoL in Arm 1A and Arm 1B using EORTC QLQ-C30 questionnaire.
  The EORTC QLQ-C30 is a 30-item, tumor-specific, patient-based questionnaire designed for self-administration. The form scores range from 0 to 100. Higher scores indicated worse symptomatic problems.
Health-related quality of life (HRQoL) by EORTC QLQ-PAN26 in Arm 1A and in Arm 1B | up to 5 years
  To assess HRQoL in Arm 1A and Arm 1B using EORTC QLQ-PAN26 questionnaire.
  The EORTC QLQ-PAN26 is a module specific to pancreatic cancer, to be used in conjunction to the EORTC QLQ-C30. It contains 26 items. As for the EORTC QLQ-C30, one score is generated for each item, in order that a high score represents a high functional level and a high symptomatic level. Estimated duration: 10 min.
6-month progression-free survival (PFS) post randomization (R1) of standard NALIRIFOX in Arm 1B | 6 months
  To assess a 6-month PFS post R1 of standard NALIRIFOX in Arm 1B

CONTACTS AND LOCATIONS:
Overall Officials: Cindy NEUZILLET, MD, Principal Investigator — Institute Curie, Versailles Saint-Quentin University, Saint-Cloud,
Locations (12):
- France (12):
  - CHU de Besançon, Besançon
  - CHU de Grenoble, La Tronche
  - CHU de Lille, Lille
  - Institut Curie, Paris
  - Pitié Salpêtrière Hospital, Paris
  - Saint-Antoine Hospital, Paris
  - CHU de Poitiers, Poitiers
  - CHU de Reims, Reims
  - Institute Curie, Saint-Cloud
  - CHU de Saint Etienne, Saint-Etienne
  - Hôpital d'Instruction des Armées Bégin, Saint-Mandé
  - Paul Brousse Hospital, Villejuif

IPD SHARING:
Plan to Share IPD: No